CLINICAL TRIAL: NCT05142735
Title: Effects of N-acetylcysteine on Psychosis-like Symptoms and a Neurophysiological Biomarker of the Clinical High Risk for Schizophrenia
Brief Title: Effects of NAC on Symptoms of CHR Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 054-2020
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Prodromal Schizophrenia
Keywords: psychosis; schizophrenia; N-acetylcysteine; prodrome; mismatch negativity; event-related potentials; clinical high risk state
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders; Schizophrenia | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of NAC or placebo groups in parallel for the duration of the study. This will be a randomized, double-blind, placebo-controlled trial.
  Participants will be randomized to take either NAC 2000 mg or placebo, in the form of oral capsules, every morning for 8 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and research staff are blinded to the conditions. Research Pharmacy staff are unblinded and responsible for randomization and NAC or placebo dispensing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): N-Acetylcysteine 2000 mg (4 x 500-mg tablets) orally every morning for 8 weeks
  Interventions: Dietary Supplement: N-Acetylcysteine
- Placebo Comparator (Placebo Comparator): N-Acetylcysteine Placebo tablet matching N-Acetylcysteine orally every morning for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: N-Acetylcysteine — 2000 mg (4 x 500-mg tablets) every morning
  Other Names: NAC
  Arms: Experimental
Dietary Supplement: Placebo — 4 placebo tablets every morning
  Arms: Placebo Comparator

SUMMARY:
Schizophrenia is a chronic debilitating psychotic disorder. Identifying persons with "clinical high-risk" (CHR) symptoms, which are like those of schizophrenia but less severe, and providing psychiatric care to these individuals has been shown to help prevent psychosis. Current medications used for CHR symptoms, however, are associated with substantial side effect burden. Therefore, practice guidelines do not recommend current medications as routine treatment for the CHR state, and there is a need to identify new treatments for this condition.

Research suggests that abnormal brain oxidative stress may contribute to schizophrenia, offering a potential novel treatment target in the CHR state. Oxidative stress is an excess of free radicals, which are generated from normal metabolism and environmental exposures, and can damage cells. Antioxidants in the body normally neutralize free radicals. Antioxidant deficiency could result in excess oxidative stress that damages brain cells, leading to schizophrenia. Recent studies suggest that N-acetylcysteine (NAC), a precursor of the most abundant brain antioxidant, glutathione, may be a safe, well-tolerated treatment for schizophrenia. In light of this, NAC may also reduce symptoms and brain abnormalities in CHR patients.

DETAILED DESCRIPTION:
The primary aim is to examine the effect of NAC on psychosis-like symptoms in CHR patients. Secondary aims are to examine the effect of NAC, in these patients, on the amplitude of the mismatch negativity (MMN), an electroencephalographic event-related potential (ERP) response to rare sounds among frequent ones; and the amplitude of the N400 semantic priming effect, an ERP response to unexpected compared to expected meaningful stimuli (e.g., words, pictures); both of which have been found to be reduced in both schizophrenia and the CHR state.

This will be a randomized, double-blind, placebo-controlled trial. Ninety CHR patients will take either NAC 2000 mg orally or placebo, daily for 8 weeks. Psychosis-like symptoms will be assessed at baseline, week 4 and week 8 using the Positive symptom score of the Scale of Psychosis-Risk Symptoms in the Structured Interview for Psychosis-Risk Syndromes. MMN amplitude and the N400 semantic priming effect will be measured at baseline and week 8. We hypothesize that patients will have more improvement in psychosis-like symptoms, and greater increases in MMN amplitudes and N400 semantic priming effects, after taking NAC vs. placebo. If we find that NAC improves psychosis-like symptoms and/or these neurophysiological biomarkers of the CHR state, this would support further research on NAC as a preventive treatment against psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. meeting Criteria of Psychosis-Risk Syndromes (COPS) criteria on the Structured Interview for Psychosis-Risk Syndromes (SIPS)
2. capacity to provide informed consent
3. if female, participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure or have been post-menopausal for at least 1 year prior to screening OR participant is of child-bearing potential and agrees to use a medically approved method of birth control for the duration of the study

Exclusion Criteria:

1. meeting criteria for any other DSM-5 diagnosis at the time of the study (except -personality disorder, nicotine use disorder, or other substance use disorder in full remission)
2. concomitant or past neurological condition
3. visual impairment which is not corrected to normal by prescription glasses history of reading disability
4. past antipsychotic treatment at a therapeutic dose
5. current treatment with a psychotropic medication except antidepressants on which the participants has been on a stable dose for at least 30 days.
6. pregnancy (as identified on self-report and/or rapid urine pregnancy test) or intent to become pregnant according to self-report
7. breastfeeding or plan to do so
8. history of kidney stones
9. current treatment with an antibiotic
10. current treatment with nitroglycerin
11. allergy to any ingredients in either the investigational product or placebo product

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in positive psychosis-like symptoms from baseline to 8 weeks | Week 0 to week 8
  Measured by the Positive symptom score of the Scale of Psychosis-Risk Symptoms, where the minimum score is 0 and the maximum score is 30, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in mismatch negativity (MMN) amplitude from baseline to 8 weeks | Week 0 to week 8
  MMN amplitude will be measured as mean voltage from 135-205 ms post-stimulus onset of the ERP waveform formed by subtracting the average for standard tones from the average for deviant tones.
Change in N400 semantic priming effect from baseline to 8 weeks | Week 0 to week 8
  N400 semantic priming effect will be measured as mean voltage from 300-500 ms post-stimulus onset of the ERP waveform formed by subtracting the average for related stimuli from the average for unrelated stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kiang, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addington J, Addington D, Abidi S, Raedler T, Remington G. Canadian Treatment Guidelines for Individuals at Clinical High Risk of Psychosis. Can J Psychiatry. 2017 Sep;62(9):656-661. doi: 10.1177/0706743717719895. Epub 2017 Jul 21. PMID 28730848
- [Background] Atkinson RJ, Michie PT, Schall U. Duration mismatch negativity and P3a in first-episode psychosis and individuals at ultra-high risk of psychosis. Biol Psychiatry. 2012 Jan 15;71(2):98-104. doi: 10.1016/j.biopsych.2011.08.023. Epub 2011 Oct 13. PMID 22000060
- [Background] Breier A, Liffick E, Hummer TA, Vohs JL, Yang Z, Mehdiyoun NF, Visco AC, Metzler E, Zhang Y, Francis MM. Effects of 12-month, double-blind N-acetyl cysteine on symptoms, cognition and brain morphology in early phase schizophrenia spectrum disorders. Schizophr Res. 2018 Sep;199:395-402. doi: 10.1016/j.schres.2018.03.012. Epub 2018 Mar 24. PMID 29588126
- [Background] Cabungcal JH, Counotte DS, Lewis E, Tejeda HA, Piantadosi P, Pollock C, Calhoon GG, Sullivan E, Presgraves E, Kil J, Hong LE, Cuenod M, Do KQ, O'Donnell P. Juvenile antioxidant treatment prevents adult deficits in a developmental model of schizophrenia. Neuron. 2014 Sep 3;83(5):1073-1084. doi: 10.1016/j.neuron.2014.07.028. Epub 2014 Aug 14. PMID 25132466
- [Background] Conus P, Seidman LJ, Fournier M, Xin L, Cleusix M, Baumann PS, Ferrari C, Cousins A, Alameda L, Gholam-Rezaee M, Golay P, Jenni R, Woo TW, Keshavan MS, Eap CB, Wojcik J, Cuenod M, Buclin T, Gruetter R, Do KQ. N-acetylcysteine in a Double-Blind Randomized Placebo-Controlled Trial: Toward Biomarker-Guided Treatment in Early Psychosis. Schizophr Bull. 2018 Feb 15;44(2):317-327. doi: 10.1093/schbul/sbx093. PMID 29462456
- [Background] Flatow J, Buckley P, Miller BJ. Meta-analysis of oxidative stress in schizophrenia. Biol Psychiatry. 2013 Sep 15;74(6):400-9. doi: 10.1016/j.biopsych.2013.03.018. Epub 2013 May 15. PMID 23683390
- [Background] Hsieh MH, Shan JC, Huang WL, Cheng WC, Chiu MJ, Jaw FS, Hwu HG, Liu CC. Auditory event-related potential of subjects with suspected pre-psychotic state and first-episode psychosis. Schizophr Res. 2012 Sep;140(1-3):243-9. doi: 10.1016/j.schres.2012.06.021. Epub 2012 Jul 10. PMID 22784684
- [Background] Jahshan C, Cadenhead KS, Rissling AJ, Kirihara K, Braff DL, Light GA. Automatic sensory information processing abnormalities across the illness course of schizophrenia. Psychol Med. 2012 Jan;42(1):85-97. doi: 10.1017/S0033291711001061. Epub 2011 Jul 11. PMID 21740622
- [Background] Kim M, Lee TH, Yoon YB, Lee TY, Kwon JS. Predicting Remission in Subjects at Clinical High Risk for Psychosis Using Mismatch Negativity. Schizophr Bull. 2018 Apr 6;44(3):575-583. doi: 10.1093/schbul/sbx102. PMID 29036493
- [Background] Lavoie S, Jack BN, Griffiths O, Ando A, Amminger P, Couroupis A, Jago A, Markulev C, McGorry PD, Nelson B, Polari A, Yuen HP, Whitford TJ. Impaired mismatch negativity to frequency deviants in individuals at ultra-high risk for psychosis, and preliminary evidence for further impairment with transition to psychosis. Schizophr Res. 2018 Jan;191:95-100. doi: 10.1016/j.schres.2017.11.005. Epub 2017 Nov 11. PMID 29132815
- [Background] Lepock JR, Ahmed S, Mizrahi R, Gerritsen CJ, Maheandiran M, Drvaric L, Bagby RM, Korostil M, Light GA, Kiang M. Relationships between cognitive event-related brain potential measures in patients at clinical high risk for psychosis. Schizophr Res. 2020 Dec;226:84-94. doi: 10.1016/j.schres.2019.01.014. Epub 2019 Jan 22. PMID 30683525
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Nagai T, Tada M, Kirihara K, Yahata N, Hashimoto R, Araki T, Kasai K. Auditory mismatch negativity and P3a in response to duration and frequency changes in the early stages of psychosis. Schizophr Res. 2013 Nov;150(2-3):547-54. doi: 10.1016/j.schres.2013.08.005. Epub 2013 Sep 6. PMID 24012461
- [Background] Perez VB, Woods SW, Roach BJ, Ford JM, McGlashan TH, Srihari VH, Mathalon DH. Automatic auditory processing deficits in schizophrenia and clinical high-risk patients: forecasting psychosis risk with mismatch negativity. Biol Psychiatry. 2014 Mar 15;75(6):459-69. doi: 10.1016/j.biopsych.2013.07.038. Epub 2013 Sep 16. PMID 24050720
- [Background] Schmidt SJ, Schultze-Lutter F, Schimmelmann BG, Maric NP, Salokangas RK, Riecher-Rossler A, van der Gaag M, Meneghelli A, Nordentoft M, Marshall M, Morrison A, Raballo A, Klosterkotter J, Ruhrmann S. EPA guidance on the early intervention in clinical high risk states of psychoses. Eur Psychiatry. 2015 Mar;30(3):388-404. doi: 10.1016/j.eurpsy.2015.01.013. Epub 2015 Mar 3. PMID 25749390
- [Background] Sepehrmanesh Z, Heidary M, Akasheh N, Akbari H, Heidary M. Therapeutic effect of adjunctive N-acetyl cysteine (NAC) on symptoms of chronic schizophrenia: A double-blind, randomized clinical trial. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Mar 2;82:289-296. doi: 10.1016/j.pnpbp.2017.11.001. Epub 2017 Nov 7. PMID 29126981
- [Background] Shaikh M, Valmaggia L, Broome MR, Dutt A, Lappin J, Day F, Woolley J, Tabraham P, Walshe M, Johns L, Fusar-Poli P, Howes O, Murray RM, McGuire P, Bramon E. Reduced mismatch negativity predates the onset of psychosis. Schizophr Res. 2012 Jan;134(1):42-8. doi: 10.1016/j.schres.2011.09.022. Epub 2011 Oct 24. PMID 22024244
- [Background] Steullet P, Cabungcal JH, Monin A, Dwir D, O'Donnell P, Cuenod M, Do KQ. Redox dysregulation, neuroinflammation, and NMDA receptor hypofunction: A "central hub" in schizophrenia pathophysiology? Schizophr Res. 2016 Sep;176(1):41-51. doi: 10.1016/j.schres.2014.06.021. Epub 2014 Jul 5. PMID 25000913
- [Background] Zheng W, Zhang QE, Cai DB, Yang XH, Qiu Y, Ungvari GS, Ng CH, Berk M, Ning YP, Xiang YT. N-acetylcysteine for major mental disorders: a systematic review and meta-analysis of randomized controlled trials. Acta Psychiatr Scand. 2018 May;137(5):391-400. doi: 10.1111/acps.12862. Epub 2018 Feb 18. PMID 29457216